CLINICAL TRIAL: NCT07336433
Title: EFS Study of the Renal Nerve Mapping/Selective Renal Denervation (msRDN) System in the Absence of Antihypertensive Medications: A Prospective, Multicentre, Single-Arm Exploratory Trial
Brief Title: SMART-IC-Pilot Study
Acronym: SMART-IC-Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SyMap Medical (Suzhou), Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMART-IC-2025
Record Dates: First submitted 2025-12-18; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hypertensive Disease
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mapping/Selective Renal Denervation (Experimental): Mapping/Selective Renal Denervation
  Interventions: Device: The SymPioneer G2 Mapping/Selective Renal Denervation Device and SyMapCath Catheter II

INTERVENTIONS:
Device: The SymPioneer G2 Mapping/Selective Renal Denervation Device and SyMapCath Catheter II — Radiofrequency ablation of renal arterial sympathetic nerves

SUMMARY:
This small-scale, proof-of-concept pilot study aims to obtain preliminary evidence of msRDN procedural safety, feasibility, and short-term efficacy in patients with hypertension without medication therapy, to adequately plan an appropriate pivotal study.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm, exploratory study enrolling 15 subjects across approximately four sites with a 6-month follow-up period. Subjects are patients with uncontrolled hypertension who receive 1-2 antihypertensive medications and have completed a minimum two-week medication wash-out period prior to enrollment, or patients with uncontrolled hypertension without medication therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Documented essential hypertension
3. Resistant or drug-intolerant hypertension, particularly in patients requiring medication reduction
4. Office BP ≥ 140/90 mmHg and < 180/110 mmHg while on a stable regimen of 1-2 antihypertensive medications for ≥ 4 weeks before consent
5. Documented daytime ASBP ≥ 135 mmHg and < 170 mmHg after 2-week washout
6. Able and willing to comply with all study procedures and follow-up visit

Exclusion Criteria:

1.Renal artery anatomy on either side, unsuitable for treatment:

1. Main renal artery diameter < 4 mm or > 8 mm
2. Main renal artery length < 25 mm
3. Single functioning kidney
4. Presence of abnormal kidney (or secreting adrenal) tumors
5. Renal artery with aneurysm
6. Pre-existing renal stent or history of renal artery angioplasty
7. Prior renal denervation procedure
8. Renal artery stenosis ≥ 50% 2.Active infection within 7 days of procedure 3.Iliac/femoral artery stenosis precluding msRDN catheter insertion 4.Type I diabetes mellitus 5.eGFR <45 mL/min/1.73 m2 (by Modification of Diet in Renal Disease formula) 6.Any history of cerebrovascular event (e.g. stroke, transient ischemic event, cerebrovascular accident) 7.Any history of severe cardiovascular event (myocardial infarction, CABG, acute heart failure requiring hospitalization (NYHA III-IV) 8.Documented confirmed episode(s) of stable or unstable angina 9.Documented repeat (> 1) hospitalization for hypertensive crisis within the prior 12 months 10.Chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea 11.Primary pulmonary hypertension 12.Documented contraindication or allergy to contrast medium not amenable to treatment 13.Limited life expectancy of < 1 year at the discretion of the Investigator 14.Known drug/alcohol dependence or inability to comply with study protocol Pregnant, breastfeeding or intend to become pregnant within 12 months -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in daytime ASBP | From baseline to 2 months after RDN
  mean change in average daytime ASBP from baseline to 2 months post-procedure.

SECONDARY OUTCOMES:
Change in office SBP | From baseline to 1, 2, 3 and 6 months after RDN
  Change in Office Systolic BP from baseline to 1 month,2 months,3 months and 6 months post-procedure;
Change in average 24-hr/Night-time Ambulatory BP(Systolic and Diastolic) | From baseline to 2 months after RDN (for both 24-hr and night-time SBP/DBP); From baseline to 2 months after RDN (for daytime DBP)
  change in Average 24-hr/Night-time Ambulatory BP(Systolic and Diastolic) from baseline to 2 months and daytime ambulatory Diastolic BP from baseline to 2 months post procedure
Change in 24-hr Ambulatory BP | From baseline to 6 months after RDN
  Change in 24-hr Ambulatory BP from baseline to 6 months post-procedure
Change in anti-hypertensive Drugs | From baseline to 1, 2, 3 and 6 months after RDN
  Change in anti-hypertensive Drugs form baseline to 1 month、2 months、3 months and 6 months post-procedure;

OTHER OUTCOMES:
Success rate of the renal interventional therapy procedure | Immediately after the procedure and at 7 days post-procedure (or prior to discharge, whichever occurs first
  The renal denervation catheter can be engaged to the correct position in renal artery, successfully performed renal nerve ablation procedure and has no related complications such as renal arterial perforation;
Success rate of clinical treatment | Immediately after the procedure and at 7 days post-procedure (or prior to discharge, whichever occurs first
  Based on succeed performance of renal interventional therapy procedure , there are no the procedure-related SAE, such as acute infection and renal dysfunction. 7 days after the procedure or at the time the patient is discharged from hospital
All-cause mortality | From baseline to 1, 2, 3 and 6 months after RDN
Severe renal dysfunction (eGFR<15mL/min/m2 or renal function replacement therapy needed) | From baseline to 6 months after RDN
Rate of new-onset renal artery stenosis assessed (stenosis > 70% ) | From baseline to 2 and 6 months after RDN
AEs, SAEs and severe cardio-cerebrovascular events | From baseline to1,3 and 6 months after RDN

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided